CLINICAL TRIAL: NCT00365794
Title: Investigator Initiated Study of the Effects of Androgen Therapy on Carbohydrate and Lipid Metabolism In Elderly Men
Brief Title: Effects of Testosterone Gel on Carbohydrate and Lipid Metabolism In Elderly Obese Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Fred Sattler, MD, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCRC Protocol 1156
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Aging; Obesity; Insulin Resistance; Hypogonadism
Keywords: Aging; Older men; Abdominal obesity; Central obesity; Insulin resistance; Low testosterone
MeSH Terms: conditions — Obesity; Insulin Resistance; Hypogonadism; Obesity, Abdominal | interventions — Testosterone

STUDY DESIGN:
Masking Description: No masking. This was an open label (un-blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Open label treatment without masking with each participant serving as his own control. Measurements are compared before and after treatment.
  Interventions: Drug: Topical testosterone gel 10 g/day

INTERVENTIONS:
Drug: Topical testosterone gel 10 g/day — Testosterone gel therapy for 20 weeks
  Other Names: Androgel

SUMMARY:
A. HYPOTHESES: In older men low testosterone levels, abdominal obesity and elevated fasting insulin who are at risk for the cardiovascular complications such as heart attack and stroke.

1. Supplemental testosterone will decrease abdominal adipose tissue and hepatic fat) and appendicular fat and intramyocellular lipid in peripheral muscles (IMCL).
2. Supplemental testosterone will improve insulin sensitivity by:

   1. Decreasing hepatic glucose output (HGO), a measure of central insulin resistance
   2. increasing peipheral glucose disposal (Rd), a measure of periperal insuln sensiivity
   3. . Improving peripheral glucose disposal (Rd) by reducing IMCL
   4. Increasing appendicular skeletal muscle mass

B. OBJECTIVES:

1. Primary Objective: To determine the effects of supplemental testosterone to achieve testosterone levels in the upper normal physiologic range on central adipose tissue (abdominal and hepatic fat) and peripheral skeletal muscle fat (appendicular fat and IMCL).
2. Secondary Objectives: To determine the effects of supplemental testosterone to achieve testosterone levels in the upper normal physiologic range:on central insulin sensitivity ( hepatic glucose output ([HGO]) and peripheral insulin sensitivity (glucose disposal (Rd)

Results of this study will provide greater understanding whether androgen therapy enhances insulin sensitivity by decreasing HGO, improving peripheral Rd and if these desired effects are achieved, whether they are due to reductions in abdominal fat or liver lipid, IMCL or effects of augmenting muscle mass per se.

Results will generate hypotheses to investigate cellular and molecular mechanisms of androgen effects in persons at risk for the Metabolic Syndrome.

DETAILED DESCRIPTION:
Study Design: This is an investigator-initiated open label, study to investigate the effects of supplemental testosterone (gel formulation) to increase testosterone levels to the upper normal range in 12 older hypogonadal (testosterone levels less than 300 ng/dL) men with abdominal obesity and elevated fasting insulin levels. Subjects will be assigned to receive 10 g of transdermal testosterone (Androgel) every morning to achieve levels in the upper normal physiologic range (similar to men in the 3rd and 4th decades) for 20 weeks.

* For the primary objective, regional adipose tissue, namely DEXA measures of abdominal and appendicular fat mass and hepatic fat, and IMCL will be quantified by 1H-spectroscopy at baseline (study week 0) and at study week 20 (completion of study therapy).
* For the secondary objective, insulin sensitivity (peripheral Rd, hepatic glucose output [HGO]) and hepatic gluconeogenesis will be measured directly during a two stage hyperinsulinemic euglycemic clamp at baseline and study week 20.
* Indirect markers of lipid (adiponectin, ApoB 100) and carbohydrate metabolism (Fasting blood sugar, HOMA-IR) at study week 10, and study week 20.

All components of the study will be conducted in the USC NIH-funded (NCRR), General Clinical Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Entry Criteria:
* Men > 60 years of age
* Total testosterone < 300 ng/dL
* Waist circumference >102 cm
* Fasting insulin level > 18 U/L

Exclusion Criteria:

* PSA > 4.1, symptoms of obstructive uropathy (AUA score > 14), unexplained prostate nodule or gland firmness
* Hematocrit > 50%
* Malignancy other than cutaneous cancers
* Sleep apnea requiring CPAP
* History of myocardial infarction, angina or stroke within the previous 6 months
* Clinical diagnosis of diabetes or FPG > 126 mg/dL
* Hypothyroidism not controlled to euthyroid levels with medication for at least 3 months
* LDL-C >160 mg/dL
* Transaminases > 1.5X ULN
* Systemic anticoagulation with warfarin
* Active progressive resistance training
* Dieting for weight loss
* Active inflammatory condition (e.g. rheumatoid arthritis)
* Use of any anabolic agent (e.g. growth hormone, testosterone precursor, anabolic steroid)or cytokine therapy in the proceeding 12 months

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-08; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred R Sattler, MD, Principal Investigator — University of Southern California
Locations (1):
- LAC-USC Medical Center GCRC, Los Angeles, California, United States

REFERENCES:
- [Result] Sattler F, He J, Chukwuneke J, Kim H, Stewart Y, Colletti P, Yarasheski K, Buchanan T. Testosterone Supplementation Improves Carbohydrate and Lipid Metabolism in Some Older Men with Abdominal Obesity. J Gerontol Geriatr Res. 2014 Jun 7;3(3):1000159. doi: 10.4172/2167-7182.1000159. PMID 25392748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were primarily recruited from 2011 to 2013 and were evaluated and studied at the University of Southern California CTSI Clinical Trials Unit. 22 subjects met all eligibility requirements and begun study therapy with testosterone gel. Two did not complete treatment. Thus, 20 completed all evaluations as planned.
Pre-assignment Details: Consenting subjects were evaluated for eligibility and had to be:
  Men 60 years-or-older, with morning testosterone <400ng/dL, waist circumference ≥102cm, and evidence of insulin resistance; HgbA1c of 5.7-6.4% [20] or HOMA-IR ≥4.0. Exclusion criteria included diabetes, PSA ≥4.0μg/L, hct ≥50%, AST ≥2X ULN, concurrent inflammatory condition.
Groups:
- Single Arm: Open label treatment with each participant serving as his own control. Data is compared before and after treatment.
  Topical testosterone (Androgel) 10 g/day: Testosterone therapy for 20 weeks
Period: Overall Study
Arm/Group | Single Arm
Started (All milestones were met 1) target number enrolled and 2) all finished study therapy and measurements) | 22 (22 subjects were enrolled since only 20 completed all post treatment measures.)
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: open label treatment with testosterone gel
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 67.5 [62.0 to 78.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
AM total testosterone level [Median (Full Range); unit: nmoles/liter] | 10.6 [5.2 to 13.9]
waist circumference [Median (Full Range); unit: centimeters] | 114 [104 to 122]
blood panels [Median (Full Range); unit: mmole/liter]
  total cholesterol | 4.61 [3.00 to 6.73]
  LDL cholesterol | 3.11 [0.98 to 5.00]
  HDL cholesterol | 1.06 [0.62 to 1.76]
  Fasting triglycerides | 1.59 [0.72 to 4.87]
Patient history at enrollment [Count of Participants; unit: Participants]
  Family history of diabetes | 4
  Smoking ever | 14
  Smoking currently | 0
  On Rx for lipid disorder | 12
  On Rx for hypertension | 10
Body compotion [Median (Full Range); unit: kilograms] — kilograms as measured by DEXA
  kilograms
    Total body mass | 104.5 [84.4 to 133.6]
    Total fat mass | 34.6 [24.3 to 57.1]
    Trunk fat mass | 19.3 [13.6 to 30.0]
    Extremity fat mass | 12.9 [9.1 to 27.6]
    Total lean body mss | 64.3 [47.1 to 75.0]
    Extremity lean mass | 29.1 [21.2 to 34.1]
Percentage of body fat [Median (Full Range); unit: percentage] | 31.5 [23.9 to 42.7]
Insulin senstivity [Median (Full Range); unit: dL/min per μU/mL;]
  Whole body insulin sensivity | 2.93 [1.07 to 8.51]
  Hepatic glucose output | 2.89 [0.03 to 7.83]
  Rate of glucose disposal | 2.93 [1.07 to 8.51]
HOMA-IR [Median (Full Range); unit: microU/L) x fasting glucose (nmol/L)/22.] | 3.55 [0.64 to 11.4]
Basal free fatty acids [Median (Full Range); unit: mEq/L] | 0.35 [0.24 to 0.53]
Change in glucose clamp free fatty acids over 0 to 4 hours [Median (Full Range); unit: grams] | 0.30 [0.17 to 0.41]
Hepatic lipid [Median (Full Range); unit: ratio] — Measurement is adjusted for water content and commonly reported as ratio
  ratio | 0.11 [0.01 to 1.13]
Intramyocellular lipid (IMCL) [Median (Full Range); unit: ratio] — IMCL is commonly adjusted for creatine (Cr) content and reported as a raio
  ratio | 5.8 [0.2 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Mass and Regional Adipose Adiposiy
Description: Change in total body mass, total fat mass, trunk fat, and extremity fat
Time Frame: Baseline to 20 weeks
Population: Data for one participant was not available
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm
Number analyzed (Participants) | 19
kilograms
  Total body mass | 0.3 [-4.8 to 4.1]
  Total fat mass | -1.4 [-7.4 to 2.0]
  Trunk fat mass | -0.9 [-4.6 to 0.2]
  Extremity fat mass | -0.7 [-3.0 to 2.3]
Statistical Analysis 1: Comparison: Single Arm; Total body mass; Test type: Other; p = 0.77, t-test, 2 sided
Statistical Analysis 2: Comparison: Single Arm; Total fat mass; Test type: Other; p = 0.003, t-test, 2 sided
Statistical Analysis 3: Comparison: Single Arm; Statistical analysis is for change in trunk fat mass after 20 weeks of testosterone gel; Test type: Other; p = 0.0007, t-test, 2 sided
Statistical Analysis 4: Comparison: Single Arm; Statistical analysis is for change in extremity fat mass after 20 weeks of testosterone gel; Test type: Other; p = 0.01, t-test, 2 sided

2. Primary Outcome: Change in Hepatic Lipid
Description: Amount of liver fat is highly predictive of insulin resistance. Hepatic fat is measured by MR spectroscopy and adjusted for H2O and results are reported as ratio of these two.
Time Frame: Baseline to week 20
Population: Data not available for one subject
Measure: Median (Full Range); unit: ratio
Arm/Group | Single Arm
Number analyzed (Participants) | 19
ratio | -36 [-84 to 127]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.12, t-test, 2 sided — No adjustment in p for multiple comparisons

3. Primary Outcome: Intramyocellular Lipid (IMCL)
Description: IMCL is quantified by MR spectroscopy of the anterior tibialis muscle of the leg. The value is adjusted for creatine and reported as a ratio
Time Frame: Baseline to week 20
Population: data not available for 5 subjects
Measure: Median (Full Range); unit: ratio
Arm/Group | Single Arm
Number analyzed (Participants) | 15
ratio | -30 [-85 to 43]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.008, t-test, 2 sided

4. Secondary Outcome: Change in Percentage of Total Body Fat
Description: Percentage of total body fat is quantified by DEXA scanning
Time Frame: Baseline and 20 weeks
Population: Data not available for one subject
Measure: Median (Full Range); unit: percentage of total body fat
Arm/Group | Single Arm
Number analyzed (Participants) | 19
percentage of total body fat | -1.6 [-6.5 to 0.1]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.0002, t-test, 2 sided — No adjustment for multiple comparisons

5. Secondary Outcome: Change in Total and Regional Carbohydrate Metabolism During a 2-hr Hyperinsulinemic Euglycemic Clamp and [6,6-2H2] Glucose Studies (Peripheral Glucose Disposal [Rd],Hepatic Glucose Output [HGO])
Description: In the final analysis, total and regional carbohydrate metabolism during a 2-hr hyperinsulinemic euglycemic clamp (peripheral glucose disposal [Rd],hepatic glucose output [HGO]) were analyzed by mass transfer of glucose during both stages of the clamp relative to insulin levels.
Time Frame: Baseline and 20 weeks
Measure: Median (Full Range); unit: dL/min per μU/mL
Arm/Group | Single Arm
Number analyzed (Participants) | 20
dL/min per μU/mL
  Whole body insulin sensitiity | 1.05 [-2.44 to 3.73]
  hepaic glucose output (HGO) | -0.16 [-2.58 to 7.49]
  peripheral glucose disposal (Rd) | 1.16 [-3.08 to 3.85]
Statistical Analysis 1: Comparison: Single Arm; Statistical analysis for change in whole body insulin sensitivity after treatment with testosterone gel for 20 weeks; Test type: Other; p = 0.04, t-test, 2 sided
Statistical Analysis 2: Comparison: Single Arm; Statistical analysis for change in hepatic glucose output (measure of central insulin sensitivity) after treatment with testosterone gel for 20 weeks; Test type: Other; p = 0.59, t-test, 2 sided
Statistical Analysis 3: Comparison: Single Arm; Statistical analysis for change in rate of peripheral glucose disposal (test of peripheral insulin sensitivity) after treatment with testosterone gel for 20 weeks; Test type: Other; p = 0.03, t-test, 2 sided

6. Secondary Outcome: Change in Skeletal Muscle Mass by DEXA
Description: Skeletal muscle mass was assesed by regional DEXA to quantify appendicular lean tissues which is primarily muscle.
Time Frame: Baselne to 20 weeks
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm
Number analyzed (Participants) | 20
kilograms | 1.2 [-1.1 to 4.8]
Statistical Analysis 1: Comparison: Single Arm; Change in DEXA extremity (appendicular) lean tissue, a measure of extremity muscle mass after 20 weeks ot treatent with testosterone gel; Test type: Other; p = 0.0006, t-test, 2 sided

7. Secondary Outcome: Plasma Lipids
Time Frame: Baseline to week 20
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Single Arm
Number analyzed (Participants) | 20
mg/dL
  Fasting triglycerides | -0.33 [-2.70 to 0.43]
  Total cholesterol | -0.52 [-1.74 to 0.88]
  LDL cholesterol | -0.23 [-1.45 to 0.70]
  HDL cholesterol | -0.10 [-0.60 to 0.05]
Statistical Analysis 1: Comparison: Single Arm; A change in 20 plasma lipids (fasting triglycerides and lipid fractions) after 20 weeks of treatment with testosterone gel; Test type: Other — Test for fasting triglycerides; p = 0.02, t-test, 2 sided
Statistical Analysis 2: Comparison: Single Arm; [analysis description as in outcome 7, analysis 1]; Test type: Other — Test for total cholesterol; p = 0.004, t-test, 2 sided
Statistical Analysis 3: Comparison: Single Arm; nts A change in 20 plasma lipids (fasting triglycerides and lipid fractions) after 20 weeks of treatment with testosterone gel; Test type: Other — Test for LDL cholesterol; p = .02, t-test, 2 sided
Statistical Analysis 4: Comparison: Single Arm; [analysis description as in outcome 7, analysis 1]; Test type: Other — Test for HDL cholesterol; p = 0.004, t-test, 2 sided

8. Secondary Outcome: Change in HOMA-IR
Description: HOMA-IR is a measure of insulin resistance
Time Frame: Baseline to week 20
Measure: Median (Full Range); unit: microU/L) x fasting glucose (nmol/L)/22
Arm/Group | Single Arm
Number analyzed (Participants) | 20
microU/L) x fasting glucose (nmol/L)/22 | -0.75 [-6.94 to 4.18]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.06, t-test, 2 sided

9. Secondary Outcome: Change in Basal FFAs in Plasma
Description: FFA (plasma free fatty acids) are measure of lipid metabolism
Time Frame: Baseline to week 20
Measure: Median (Full Range); unit: mEq/L
Arm/Group | Single Arm
Number analyzed (Participants) | 20
mEq/L | -0.1 [-0.22 to 0.21]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.97, t-test, 2 sided

10. Secondary Outcome: Change in Plasma Free Fatty Acids During Glucose Clamp
Time Frame: Baseline to 20 weeks
Measure: Median (Full Range); unit: grams
Arm/Group | Single Arm
Number analyzed (Participants) | 20
grams | -0.1 [-0.12 to 0.17]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.83, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 20 weeks for each participant
Description: No serious adverse events occurred.
Groups:
- Open Label Testosterone Treatment: No serious adverse events occurred
  PSA and Framingham CV Disease Risk Score did not increase
Arm/Group | Open Label Testosterone Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Testosterone Treatment (N=20)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary limitation of this small pilot study is that it does not have a control group.

It is also likely under-powered and thus unable to show significance differences for some measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No